CLINICAL TRIAL: NCT00001150
Title: Induction of Suction Blisters in Patients With Urticaria, Blistering Diseases, Inflammatory Dermatoses and Neoplastic Disorders, and in Normal Volunteers
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 760293; 76-C-0293
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-03

CONDITIONS: Dermatitis; Healthy; Neoplasm; Urticaria; Vesiculobullous Skin Disease
Keywords: Blister Formation; Inflammatory Mediator Assay; Ultraviolet Radiation
MeSH Terms: conditions — Dermatitis; Neoplasms; Urticaria; Skin Diseases, Vesiculobullous

SUMMARY:
The use of a suction blister apparatus has facilitated study of the immunologic capacity of human epidermal cells. We have been able to prepare purified populations of these cells after blister formation. Specifically, using the blister tops, we are able to enrich for epidermal Langerhans cells which are very potent stimulators in antigen presenting assays. Thus, this normal volunteer study provides an important source of fresh epidermal tissue from which we can study normal epidermal Langerhans cell function. In addition, we have recently used blister roofs in important experimental models of HIV-1 transmission. There is no other method available for assessing the biologic function of freshly isolated Langerhans cells without altering their milieu. It is a very safe and effective way to obtain human epidermal samples.

DETAILED DESCRIPTION:
The use of a suction blister apparatus has facilitated study of the immunologic capacity of human epidermal cells. We have been able to prepare purified populations of these cells after blister formation. Specifically, using the blister tops, we are able to enrich for epidermal Langerhans cells which are very potent stimulators in antigen presenting assays. Thus, this normal volunteer study provides an important source of fresh epidermal tissue from which we can study normal epidermal Langerhans cell function. In addition, we have recently used blister roofs in important experimental models of HIV-1 transmission. There is no other method available for assessing the biologic function of freshly isolated Langerhans cells without altering their milieu. It is a very safe and effective way to obtain human epidermal samples.

ELIGIBILITY:
INCLUSION CRITERIA

Patients with urticaria of all types, blistering diseases, inflammatory dermatoses and neoplastic skin diseases.

Patients 18 years of age or older.

No pregnant women.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2000
Dates: Start 1976-10; Study Completion 2004-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Blauvelt A, Clerici M, Lucey DR, Steinberg SM, Yarchoan R, Walker R, Shearer GM, Katz SI. Functional studies of epidermal Langerhans cells and blood monocytes in HIV-infected persons. J Immunol. 1995 Apr 1;154(7):3506-15. PMID 7897231
- [Background] Blauvelt A, Chougnet C, Shearer GM, Katz SI. Modulation of T cell responses to recall antigens presented by Langerhans cells in HIV-discordant identical twins by anti-interleukin (IL)-10 antibodies and IL-12. J Clin Invest. 1996 Mar 15;97(6):1550-5. doi: 10.1172/JCI118578. PMID 8617889
- [Background] Zaitseva M, Blauvelt A, Lee S, Lapham CK, Klaus-Kovtun V, Mostowski H, Manischewitz J, Golding H. Expression and function of CCR5 and CXCR4 on human Langerhans cells and macrophages: implications for HIV primary infection. Nat Med. 1997 Dec;3(12):1369-75. doi: 10.1038/nm1297-1369. PMID 9396607